CLINICAL TRIAL: NCT00001921
Title: Integrating EEG/MEG and fMRI: Activity Correlation Between Frontal and Temporal Lobe Structures in Schizophrenic Patients, Their Siblings and Unrelated Normal Volunteers
Brief Title: Electrophysiology and Blood Flow in Patients With Schizophrenia and Their Siblings
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990172; 99-M-0172
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2018-06-08

CONDITIONS: Healthy; Schizophrenia
Keywords: Functional Connectivity; Frontotemporal Interaction; Electrophysiology; Functional Magnetic Resonance Imaging; Healthy Subjects; Schizophrenia; MEG; Neuroimaging; EEG; MRI
MeSH Terms: conditions — Schizophrenia

SUMMARY:
This study will explore how the brain works during memory testing in an effort to understand why some patients with schizophrenia have memory difficulties.

Patients with schizophrenia and their unaffected family members are eligible for this study. Studying family members may help identify the genes related to the memory deficit in schizophrenia. Normal volunteers will also be studied.

Normal volunteers, patients with schizophrenia, and their family members interested in participating in this study will be screened with a complete medical examination and psychiatric assessment, and performance of simple tasks. Study participants will be shown numbers on a screen and asked to recall them after a brief period. This will be done during electroencephalographic (EEG) recording, in which electrodes attached to the scalp measure the brain s electrical activity. The same test will be repeated while the patient has magnetic resonance imaging of the brain. The combined MRI and EEG testing will permit better localization of the brain s electrical activity.

...

DETAILED DESCRIPTION:
It is the aim of this study to investigate the functional activation and coupling between brain regions in normals, patients with schizophrenia and unaffected family members. We will perform electrophysiological recordings (MEG, EEG) during cognitive activation (Continuous Performance Task, Sternberg paradigm, working memory). We will focus on the investigation of oscillatory brain activity as this is considered to be crucial for information processing related to neuronal integration. The measurements will be closely adapted to equivalent fMRI-measurements presented as an independent protocol (00-M-0085). The combination of both methods will help to improve activity source localization (MEG/EEG) and correlation of this activity between different parts of the brain. In addition, local activity patterns (fMRI) can be better characterized in the time domain (tonic versus phasic BOLD-activation). We will address whether cognitive activation goes along with an increase or decrease of correlation between regional brain areas. In this context, we will investigate whether this correlated activation pattern is different in schizophrenics and unaffected siblings when compared with normals. The study is integrated with the schizophrenia-sibling study (95-M-0150). Siblings of schizophrenic patients are investigated in order to achieve a better understanding of the genetic determination of schizophrenia-related pathophysiology.

ELIGIBILITY:
* INCLUSION CRITERIA:

Controls:

1. No psychiatric or severe chronic medical illness at the time of the study, and by history. This includes the absence of substance abuse histories, learning disabilities and all DSM IV disorders. The investigators will evaluate medical histories and medical conditions that are judged not to interfere with the study may be allowed.
2. No use of psychotropic substances in the last 3 months.
3. There is no upper age limit the lower age limit is 18 years.

Patients:

1) Schizophrenia, any subtype or schizoaffective disorder according to DSM IV, as detailed in protocol # 89-M-0160 ("Inpatient evaluation of neuropsychiatric inpatients", Dr. Jose Apud, principal investigator) and # 95-M-0150 ("A Longitudinal Investigation of Siblings of Schizophrenic and Manic-Depressive Patients", Dr. Daniel R. Weinberger, principal investigator).

EXCLUSION CRITERIA:

Controls and patients:

1. Impaired hearing.
2. Pregnancy (only for purpose of MRI procedures under separate protocols)
3. Head trauma with loss of consciousness in the last year or any evidence of functional impairment due to and persisting after head trauma. Patients or healthy volunteers with a known risk from exposure to high magnetic fields (e.g. patients with pace makers) and those who have metallic implants (e.g. braces) in the head region (likely to create artifact on the MRI scans) will be excluded from participating in the fMRI studies.

Patients:

1. Coexistence of another major mental illness at the time of the study. If the patients experienced other mental illnesses in the past (e.g. a learning disability or major depression), then this should be judged to be fully recovered.
2. Criteria for substance abuse met in the last 6 months.
3. Criteria for substance dependence met in the last year. If criteria for dependence were met in the past, then the duration of the disorder was less than 3 years, or not judged to have produced long-term brain changes to allow the patient to be in the study.
4. Major concurrent medical illness likely to interfere with the acquisition of the task.
5. Concomitant medications which could interfere with performance on the task.
6. Presence of dyskinetic movements of the face and tongue (likely to interfere with eyeblink measures), or of gross involuntary movements of the whole body (likely to interfere with positioning in the MRI scanner).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1386 (Actual)
Dates: Start 1999-09-21; Study Completion 2018-06-08

CONTACTS AND LOCATIONS:
Overall Officials: Karen F Berman, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rutter L, Nadar SR, Holroyd T, Carver FW, Apud J, Weinberger DR, Coppola R. Graph theoretical analysis of resting magnetoencephalographic functional connectivity networks. Front Comput Neurosci. 2013 Jul 12;7:93. doi: 10.3389/fncom.2013.00093. eCollection 2013. PMID 23874288
- [Background] Siebenhuhner F, Weiss SA, Coppola R, Weinberger DR, Bassett DS. Intra- and inter-frequency brain network structure in health and schizophrenia. PLoS One. 2013 Aug 26;8(8):e72351. doi: 10.1371/journal.pone.0072351. eCollection 2013. PMID 23991097
- [Background] Altamura M, Carver FW, Elvevag B, Weinberger DR, Coppola R. Dynamic cortical involvement in implicit anticipation during statistical learning. Neurosci Lett. 2014 Jan 13;558:73-7. doi: 10.1016/j.neulet.2013.09.043. Epub 2013 Sep 27. PMID 24080375
- [Derived] Rubinstein DY, Eisenberg DP, Carver FW, Holroyd T, Apud JA, Coppola R, Berman KF. Spatiotemporal Alterations in Working Memory-Related Beta Band Neuromagnetic Activity of Patients With Schizophrenia On and Off Antipsychotic Medication: Investigation With MEG. Schizophr Bull. 2023 May 3;49(3):669-678. doi: 10.1093/schbul/sbac178. PMID 36772948